CLINICAL TRIAL: NCT06399783
Title: Topical Simvastatin Versus Topical Steroid in Treatment of Alopecia Areata: Clinical, Dermoscopic and Immunohistochemical Study
Brief Title: Topical Simvastatin Versus Topical Steroid in Treatment of Alopecia Areata
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Alaa Gamal Ahmed Makhlouf, Principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Sim vs Cs
Record Dates: First submitted 2024-05-01; First posted 2024-05-06 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Alopecia Areata
MeSH Terms: conditions — Alopecia Areata | interventions — Simvastatin; Mometasone Furoate

STUDY DESIGN:
Intervention Model Description: Patients will be divided randomly into three groups:
  Group A: Patients will be treated by topical application of simvastatin cubosomal nanoparticled twice daily for 6 months.
  Group B: Patients will be treated by fractional CO2 laser for 6 sessions sessions each will be followed immediately by topical application of topical simvastatin.
  Group C: Patients will be treated by fractional CO2 laser for 6 sessions each will be followed immediately by topical application of topical steroid.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Simvastatin — Group of patients will be treated by topical application of simvastatin cubosomal nanoparticled twice daily for 6 months, while another group will be treated by fractional CO2 laser for 6 sessions sessions each will be followed immediately by topical application of topical simvastatin.
Drug: Mometasone Furoate — Patients will be treated by fractional CO2 laser for 6 sessions each will be followed immediately by topical application of Mometasone Furoate.
Procedure: Fractional CO2 laser — Fractional CO2 laser will be used for assisted drug delivery for both topical simvastatin and mometasone Furoate.

SUMMARY:
Alopecia areata (AA) is an autoimmune disorder characterized by non-scarring hair loss of the scalp or any hair-bearing surface.

Alopecia areata affects approximately 2% of the general population. AA has a significant influence on patients' quality of life and may induce psychological disorders.

In AA, CD4+ and CD8+ T-cells violate the immune privilege of the anagen hair follicle, leading to loss of the growing hair shaft. A genome-wide association study demonstrated a genetic predisposition to AA . Additionally, environmental insults, such as viral infections, trauma, or psychosocial stress, have also been suspected to possibly contribute to the development of the disease .

The clinical manifestations of AA vary from small well-defined patches of hair loss to the diffuse involvement of the scalp or the entire body. The majority of AA patients experience unpredictable relapsing and remitting episodes. In a number of patients, it can be persistent, especially when the hair loss is extensive.

DETAILED DESCRIPTION:
There are many treatment modalities for AA including topical treatment, intralesional injections, systemic corticosteroids, systemic immunosuppressants like methotrexate or cyclosporine, excimer laser and photochemotherapy . To date, the majority of traditional treatments for AA are of limited efficacy with a high risk of adverse effects .

Topical corticosteroids are widely used in the treatment of limited patchy AA and as a first-line therapy for children. They are also recommended as an adjunctive therapy to systemic treatments in more severe forms .

Statins are well known lipid-lowering medications. They have anti-inflammatory and immunomodulatory effects. Simvastatin belongs to the statin family. Lately, Simvastatin is utilized in treatment of several dermatological diseases . It showed efficacy in treatment of psoriasis, vitiligo, xanthomas , atopic dermatitis and acne vulgaris.

In several case reports, AA patients were successfully treated with systemic simvastatin . DelCanto, 2020 studied the effect of topical simvastatin in animal model of AA and concluded that it induced hair re-growth, suggesting that it could be a new efficient therapy for AA.

Statins are theorized to induce hair regrowth in AA by inhibiting signal transducers and activators of transcription (STAT) phosphorylation that activates several important inflammatory cytokines and also by altering the balance of Th1/Th2, suppressing IL-17, and inhibiting lymphocyte migration.

Fractional laser has been reported to be successful in treating AA. Fractional CO2 laser is assumed to help in treatment of AA through stimulation of T-cell apoptosis, arrest of hair follicles in the telogen stage, and promotion of the anagen stage. Also, Fractional CO2 laser creates microchannels in the epidermis to improve drug delivery into the skin.

ELIGIBILITY:
Inclusion Criteria:

* Patients with patchy alopecia areata involving < 50% of the total scalp.

Exclusion Criteria:

* Alopecia totalis and alopecia universalis.
* Cicatricial alopecia.
* Other causes of hair loss such as; endocrine or immunological disease.
* Skin disease in the affected area.
* Hypersensitivity or allergy to any of the treatment products used.
* Patient using treatment (topical or systemic) for alopecia areata in the last 2 months.
* Pregnant and lactating females.
* Patients with history of hypertrophic scars or keloid formation.
* Patients with active infection at the site of the lesion.

Ages: 6 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 54 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of hair regrowth in alopecia areata using SALT score. | 24 weeks
  The scalp is divided into four parts on the basis of surface area as follows: vertex or top = 40% (0.40), right side = 18% (0.18), left side = 18% (0.18) and the posterior aspect = 24% (0.24). Percentage of hair loss in any of the four areas is multiplied by the percentage of the scalp covered in that area. The SALT score is the sum of the percentage of hair loss in all the areas mentioned above.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Adami M, Prudente Ada S, Mendes DA, Horinouchi CD, Cabrini DA, Otuki MF. Simvastatin ointment, a new treatment for skin inflammatory conditions. J Dermatol Sci. 2012 May;66(2):127-35. doi: 10.1016/j.jdermsci.2012.02.015. Epub 2012 Mar 3. PMID 22455735
- [Background] Ahmadvand A, Yazdanfar A, Yasrebifar F, Mohammadi Y, Mahjub R, Mehrpooya M. Evaluating the Effects of Oral and Topical Simvastatin in the Treatment of Acne Vulgaris: A Double-blind, Randomized, Placebo-controlled Clinical Trial. Curr Clin Pharmacol. 2018;13(4):279-283. doi: 10.2174/1574884713666180821143545. PMID 30129417
- [Background] Al Salman M, Ghiasi M, Farid AS, Taraz M, Azizpour A, Mahmoudi H. Oral simvastatin combined with narrowband UVB for the treatment of psoriasis: A randomized controlled trial. Dermatol Ther. 2021 Sep;34(5):e15075. doi: 10.1111/dth.15075. Epub 2021 Aug 19. PMID 34327798
- [Background] Cervantes J, Jimenez JJ, DelCanto GM, Tosti A. Treatment of Alopecia Areata with Simvastatin/Ezetimibe. J Investig Dermatol Symp Proc. 2018 Jan;19(1):S25-S31. doi: 10.1016/j.jisp.2017.10.013. PMID 29273101
- [Background] Cheung K, Powers EM, McKillip J, Powers JG. Effect of statin use on incidence of eczema and atopic dermatitis: A retrospective cohort study. J Am Acad Dermatol. 2021 Feb;84(2):534-535. doi: 10.1016/j.jaad.2020.05.015. Epub 2020 May 11. No abstract available. PMID 32407738
- [Background] Childs JM, Sperling LC. Histopathology of scarring and nonscarring hair loss. Dermatol Clin. 2013 Jan;31(1):43-56. doi: 10.1016/j.det.2012.08.001. Epub 2012 Sep 26. PMID 23159175
- [Background] Cho S, Choi MJ, Zheng Z, Goo B, Kim DY, Cho SB. Clinical effects of non-ablative and ablative fractional lasers on various hair disorders: a case series of 17 patients. J Cosmet Laser Ther. 2013 Apr;15(2):74-9. doi: 10.3109/14764172.2013.764436. Epub 2013 Mar 6. PMID 23464363
- [Background] Choi JW, Suh DW, Lew BL, Sim WY. Simvastatin/Ezetimibe Therapy for Recalcitrant Alopecia Areata: An Open Prospective Study of 14 Patients. Ann Dermatol. 2017 Dec;29(6):755-760. doi: 10.5021/ad.2017.29.6.755. Epub 2017 Oct 30. PMID 29200765
- [Background] El-Husseiny R, Elframawy S, Abdallah M. Comparative study between fractional carbon dioxide laser vs intralesional steroid injection in treatment of alopecia areata. Dermatol Ther. 2020 Jul;33(4):e13742. doi: 10.1111/dth.13742. Epub 2020 Jul 9. PMID 32478930
- [Background] Islam N, Leung PS, Huntley AC, Gershwin ME. The autoimmune basis of alopecia areata: a comprehensive review. Autoimmun Rev. 2015 Feb;14(2):81-9. doi: 10.1016/j.autrev.2014.10.014. Epub 2014 Oct 12. PMID 25315746
- [Background] Issa MC, Pires M, Silveira P, Xavier de Brito E, Sasajima C. Transepidermal drug delivery: a new treatment option for areata alopecia? J Cosmet Laser Ther. 2015 Feb;17(1):37-40. doi: 10.3109/14764172.2014.967778. Epub 2014 Oct 16. PMID 25260052
- [Background] Karimkhani C, Boyers LN, Prescott L, Welch V, Delamere FM, Nasser M, Zaveri A, Hay RJ, Vos T, Murray CJ, Margolis DJ, Hilton J, MacLehose H, Williams HC, Dellavalle RP. Global burden of skin disease as reflected in Cochrane Database of Systematic Reviews. JAMA Dermatol. 2014 Sep;150(9):945-51. doi: 10.1001/jamadermatol.2014.709. PMID 24807687
- [Background] Lattouf C, Jimenez JJ, Tosti A, Miteva M, Wikramanayake TC, Kittles C, Herskovitz I, Handler MZ, Fabbrocini G, Schachner LA. Treatment of alopecia areata with simvastatin/ezetimibe. J Am Acad Dermatol. 2015 Feb;72(2):359-61. doi: 10.1016/j.jaad.2014.11.006. No abstract available. PMID 25592347
- [Background] Lee HH, Gwillim E, Patel KR, Hua T, Rastogi S, Ibler E, Silverberg JI. Epidemiology of alopecia areata, ophiasis, totalis, and universalis: A systematic review and meta-analysis. J Am Acad Dermatol. 2020 Mar;82(3):675-682. doi: 10.1016/j.jaad.2019.08.032. Epub 2019 Aug 19. PMID 31437543
- [Background] Li A, Meng X, Xing X, Tan H, Liu J, Li C. Efficacy and Influence Factors of 308-nm Excimer Lamp with Minoxidil in the Treatment of Alopecia Areata. Lasers Surg Med. 2020 Oct;52(8):761-767. doi: 10.1002/lsm.23210. Epub 2020 Jan 9. PMID 31919885
- [Background] Meah N, Wall D, York K, Bhoyrul B, Bokhari L, Sigall DA, Bergfeld WF, Betz RC, Blume-Peytavi U, Callender V, Chitreddy V, Combalia A, Cotsarelis G, Craiglow B, Donovan J, Eisman S, Farrant P, Green J, Grimalt R, Harries M, Hordinsky M, Irvine AD, Itami S, Jolliffe V, King B, Lee WS, McMichael A, Messenger A, Mirmirani P, Olsen E, Orlow SJ, Piraccini BM, Rakowska A, Reygagne P, Roberts JL, Rudnicka L, Shapiro J, Sharma P, Tosti A, Vogt A, Wade M, Yip L, Zlotogorski A, Sinclair R. The Alopecia Areata Consensus of Experts (ACE) study: Results of an international expert opinion on treatments for alopecia areata. J Am Acad Dermatol. 2020 Jul;83(1):123-130. doi: 10.1016/j.jaad.2020.03.004. Epub 2020 Mar 9. PMID 32165196
- [Background] Meguid AMA, Ghazally A, Ahmed AM, Bakr RM. Fractional carbon dioxide laser alone and as an assisted drug delivery for treatment of alopecia areata: a clinical, dermoscopic and immunohistochemical study. Arch Dermatol Res. 2023 Aug;315(6):1675-1688. doi: 10.1007/s00403-023-02565-x. Epub 2023 Feb 21. PMID 36809409
- [Background] Olsen EA. Investigative guidelines for alopecia areata. Dermatol Ther. 2011 May-Jun;24(3):311-9. doi: 10.1111/j.1529-8019.2011.01415.x. PMID 21689240
- [Background] Petukhova L, Duvic M, Hordinsky M, Norris D, Price V, Shimomura Y, Kim H, Singh P, Lee A, Chen WV, Meyer KC, Paus R, Jahoda CA, Amos CI, Gregersen PK, Christiano AM. Genome-wide association study in alopecia areata implicates both innate and adaptive immunity. Nature. 2010 Jul 1;466(7302):113-7. doi: 10.1038/nature09114. PMID 20596022
- [Background] Pratt CH, King LE Jr, Messenger AG, Christiano AM, Sundberg JP. Alopecia areata. Nat Rev Dis Primers. 2017 Mar 16;3:17011. doi: 10.1038/nrdp.2017.11. PMID 28300084
- [Background] Shin JM, Jung KE, Yim SH, Rao B, Hong D, Seo YJ, Kim CD, Lee Y. Putative therapeutic mechanisms of simvastatin in the treatment of alopecia areata. J Am Acad Dermatol. 2021 Mar;84(3):782-784. doi: 10.1016/j.jaad.2020.03.102. Epub 2020 Apr 9. No abstract available. PMID 32278796
- [Background] Tajiri K, Shimojo N, Sakai S, Machino-Ohtsuka T, Imanaka-Yoshida K, Hiroe M, Tsujimura Y, Kimura T, Sato A, Yasutomi Y, Aonuma K. Pitavastatin regulates helper T-cell differentiation and ameliorates autoimmune myocarditis in mice. Cardiovasc Drugs Ther. 2013 Oct;27(5):413-24. doi: 10.1007/s10557-013-6464-y. PMID 23722419
- [Background] Toussi A, Barton VR, Le ST, Agbai ON, Kiuru M. Psychosocial and psychiatric comorbidities and health-related quality of life in alopecia areata: A systematic review. J Am Acad Dermatol. 2021 Jul;85(1):162-175. doi: 10.1016/j.jaad.2020.06.047. Epub 2020 Jun 17. PMID 32561373
- [Background] Verma D, Hussain K, Namiq KS, Firoz A, Bouchama M, Raza M, Haris M, Khan S. Vitiligo: The Association With Metabolic Syndrome and the Role of Simvastatin as an Immunomodulator. Cureus. 2021 Mar 22;13(3):e14029. doi: 10.7759/cureus.14029. PMID 33898117
- [Background] Yadav D, Khandpur S, Ramam M, Singh MK, Sharma VK. Utility of Horizontal Sections of Scalp Biopsies in Differentiating between Androgenetic Alopecia and Alopecia Areata. Dermatology. 2018;234(3-4):137-147. doi: 10.1159/000490459. Epub 2018 Aug 9. PMID 30092597
- [Background] Zha S, Yu X, Wang X, Gu Y, Tan Y, Lu Y, Yao Z. Topical Simvastatin Improves Lesions of Diffuse Normolipemic Plane Xanthoma by Inhibiting Foam Cell Pyroptosis. Front Immunol. 2022 May 10;13:865704. doi: 10.3389/fimmu.2022.865704. eCollection 2022. PMID 35619689